CLINICAL TRIAL: NCT06329687
Title: A Phase 4, Single-Center, Open-Label Study Evaluating the Safety of the Tyrvaya Nasal Pump
Brief Title: A Study Evaluating the Safety of the Nasal Pump
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Internal strategy change. Not related to safety concerns.
Sponsor: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPP-010
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-03

CONDITIONS: Dry Eye; Kerato Conjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nasal Pump (Experimental): Tyrvaya nasal pump with additional silicone lubricant
  Interventions: Drug: Tyrvaya Nasal Pump

INTERVENTIONS:
Drug: Tyrvaya Nasal Pump — Tyrvaya Nasal Pump with Silicone Lubricant

SUMMARY:
The objective of this study is to determine the safety of the Tyrvaya nasal pump.

DETAILED DESCRIPTION:
The study is testing the hypothesis that the use of the Tyrvaya nasal pump with silicone lubricant does not introduce any additional safety concerns as compared to the safety of the Tyrvaya nasal pump without the additional silicone lubricant.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Have provided verbal and written informed consent
* Willing to comply with all study related visits and procedures

Exclusion Criteria:

* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- United States, California, Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nasal Pump
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nasal Pump
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events with the nasal pump with additional silicone lubricant
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Pump
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Time Frame: AE collection will start following the first administration of Tyrvaya® with additional silicone lubricant until the last follow up visit of the study at 7 days.
Description: The safety population will include all enrolled subjects who received at least one Tyrvaya ®administered with the additional silicone lubricant.
Arm/Group | Nasal Pump
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nasal Pump (N=5)
Instillation Site Irritation (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT06329687/Prot_SAP_000.pdf